CLINICAL TRIAL: NCT06008990
Title: Maternal Brain Imaging in Opioid Use Disorder
Status: Active, not recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rupa Radhakrishnan, Associate Professor of Radiology & Imaging Sciences, Indiana University
Other Study IDs: RADY-IIR-19466; 1R03DA056797-01A1 (NIH)
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder; Substance-Related Disorders; Substance Use; Pregnancy Related; Narcotic-Related Disorders; Buprenorphine Dependence
Keywords: Pregnant with Opioid Use Disorder; Opioid Use Disorder; Subutex; Buprenorphine; Pregnant taking buprenorphine/subutex
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Narcotic-Related Disorders | interventions — Buprenorphine; Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biosamples:
  During the MRI visit blood samples will be collected to estimate steady-state plasma level of buprenorphine using a population pharmacokinetic approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Mothers with Opioid Use Disorder: Planned recruitment of 20 mothers with Opioid Use Disorder who are on Buprenorphine at the time of screening.
  Interventions: Drug: Buprenorphine; Diagnostic Test: Maternal Brain MRI; Other: Blood Samples; Behavioral: Questionnaires
- Pregnant Mothers: Planned recruitment of 20 mothers who do not have any history of opioid use disorder.
  Interventions: Diagnostic Test: Maternal Brain MRI; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Buprenorphine — Pregnant mother must be taking Buprenorphine
  Groups: Pregnant Mothers with Opioid Use Disorder
Diagnostic Test: Maternal Brain MRI — Maternal Brain MRI obtained between 24-32 week gestation
Other: Blood Samples — During the MRI visit blood samples will be drawn: one hour prior to MRI, immediately before MRI, and one hour post MRI to test for Buprenorphine levels.
  Groups: Pregnant Mothers with Opioid Use Disorder
Behavioral: Questionnaires — Participants will answer questionnaires about their medical history, pregnancy, and substance use.

SUMMARY:
This research study aims to learn more about opioid use disorder (OUD) during pregnancy and how outcomes for pregnant women and their newborns can be improved. During pregnancy, people with OUD are prescribed medication-assisted therapy (MAT). The investigators are interested to know how the medication is broken down by the body during pregnancy and how effective it is. The investigators also want to learn if this medication and OUD have any effect on the different parts of the brain when compared to mothers without OUD.

ELIGIBILITY:
Pregnant Women with OUD

Inclusion Criteria:

* Age: >18 years old
* Any subject that is currently on Buprenorphine at time of screening
* Singleton pregnancy

Exclusion Criteria:

* Serious maternal medical illness
* HIV or AIDs
* Polysubstance use
* Score >9 on the PHQ-9, and score >0 on item 9 which is about suicidality
* Score of 8 or more on GAD-7
* Any contraindications for MRI
* Known or suspected major fetal congenital abnormalities

Pregnant Women with no history of OUD

Inclusion:

* Age: >18 years old
* Singleton pregnancy

Exclusion:

* Serious maternal medical illness
* HIV or AIDS
* Score of >9 on the PHQ-9, and a score of >0 on item 9 which is about suicidality
* Score of 8 or more on GAD-7
* Known or suspected major fetal congenital abnormalities
* Any contraindications for MRI
* Opioid or polysubstance abuse as identified on urine screening

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any woman of the age of 18 or older that is having a single pregnancy, and currently taking buprenorphine for opioid use disorder.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Identify alterations in Default mode network connectivity in women with prenatal opioid use disorder compares to control pregnant women without OUD on maternal brain MRI. | During MRI visit between 24-32 weeks gestational age

SECONDARY OUTCOMES:
Correlate alteration in brain rs-fMRI default mode network connectivity with steady state plasma buprenorphine exposure in pregnant women with OUD | During MRI visit between 24-32 weeks gestational age

OTHER OUTCOMES:
Assess differences in brain gray matter volumes in pregnant women with OUD compared to pregnant women without OUD. | During MRI visit between 24-32 weeks gestational age
Assess differences in brain white matter microstructure on Diffusion Tensor Imaging (DTI) in pregnant women with OUD compared to pregnant women without OUD. | During MRI visit between 24-32 weeks gestational age
Correlate alterations in brain gray matter volume and DTI metrics with steady state plasma buprenorphine exposure in pregnant women with OUD | During MRI visit between 24-32 weeks gestational age

CONTACTS AND LOCATIONS:
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided